CLINICAL TRIAL: NCT03748537
Title: Mitochondrial Function in Septic Patients
Acronym: MtiSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Borwon Wittayachamnankul, Assistant Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EME-2559-04262
Record Dates: First submitted 2018-01-23; First posted 2018-11-21 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Eligible patients for aim#3 will be randomly assigned in a 1:1 ratio of hydrocortisone and no hydrocortisone administration (control group), in a block of four patterns. Serum cortisol will be collected before administration.
  Hydrocortisone will be administered intravenously at 200 mg every 24 hours for 5 days, then tapered to a 50 mg intravenous bolus every 12 hours for days 6 to 8 and 50 mg every 24 hours for days 9 to 11, and then stopped. In control group, patient will not receive any corticosteroids for seven day after inclusion.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocortisone (Experimental): Hydrocortisone will be administered intravenously at 200 mg every 24 hours for 5 days, then tapered to a 50 mg intravenous bolus every 12 hours for days 6 to 8 and 50 mg every 24 hours for days 9 to 11, and then stopped.
  Interventions: Drug: Hydrocortisone
- No Hydrocortisone (No Intervention): In control group, patient will not receive any corticosteroids for seven day after inclusion.

INTERVENTIONS:
Drug: Hydrocortisone — After resuscitation, hypoperfusion in the sepsis patients will be treated by fluid resuscitation and vasopressor. Some groups of patients may be not responsive to this treatment (MAP <65 mmHg), administration of steroids to this group will be blindly randomized (treatment and control group). During resuscitation of septic shock patients with fluid resuscitation and vasopressors, some may not respond to treatment (MAP < 65 mmHg). Patients who have shock refractory to fluid resuscitation and norepinephrine therapy for more than 0.5 mcg/kg/min will be blindly randomized to receive steroid (treatment group) or placebo (control group). Blood samples will be obtained to determine mitochondrial functioning before, at day 1 and day 7 after administration of study medications in both groups.
  Other Names: Cortisol
  Arms: Hydrocortisone

SUMMARY:
Aim #1 To investigate the prevalence, risk and correlation of the level of sepsis with mitochondrial dysfunction in sepsis patients Aim 1.1 To investigate the prevalence of mitochondria dysfunction among sepsis patients Aim 1.2 To investigate the risk associated with mitochondrial dysfunction in sepsis patients.

Aim 1.3 To investigate the association between sepsis severity (SOFA scoring system) and the degree of mitochondrial dysfunction Aim #2 To investigate the association of mitochondrial dysfunction in sepsis with ScvO2, lactate and ∆PCO2 Aim 3.1 To investigate the therapeutic efficacy of steroids on the improvement mitochondrial function in sepsis patients Aim 3.2. To investigate the efficacy of steroids on the reduction mortality rate in sepsis patients with norepinephrine-resistant hypotension

DETAILED DESCRIPTION:
Aim #1 To investigate the prevalence, risk and correlation of the level of sepsis with mitochondrial dysfunction in sepsis patients Aim 1.1 To investigate the prevalence of mitochondria dysfunction among sepsis patients Hypothesis: Most of sepsis patients are affected by mitochondria dysfunction. Since there are many suspected cases of sepsis in the emergency department, mitochondrial function measurements will be collected. After the patients are diagnosed, the degree of mitochondrial function will be reported as a percent among all of sepsis patients.

Aim 1.2 To investigate the risk associated with mitochondrial dysfunction in sepsis patients.

Hypothesis: Some risks other than infection are associated with mitochondrial dysfunction in septic patient.

Since there are many suspected cases of sepsis in the emergency department, mitochondrial function measurements will be collected. After the patients are diagnosed, the degree of mitochondrial function will be reported at intervals. Additionally, the correlation among sex, age, obesity, underlying symptoms, cause of infection, pathogen, onset of fever before emergency department visit, number of organ dysfunction, presence of shock and other hemodynamic parameter will be collected.

Aim 1.3 To investigate the association between sepsis severity (SOFA scoring system) and the degree of mitochondrial dysfunction Hypothesis: The severity of sepsis and organ dysfunction are associated with the severity of mitochondrial dysfunction.

Since there are many suspected cases of sepsis in the emergency department, mitochondrial function measurements will be collected. After the patients are diagnosed, the degree of mitochondrial function will be reported at intervals along with the correlation with the severity of sepsis in SOFA scoring system.

Aim #2 To investigate the association of mitochondrial dysfunction in sepsis with ScvO2, lactate and ∆PCO2 Hypothesis: Persistence of high lactate and extreme change of ScvO2 or ∆PCO2 after sepsis bundle care are associated with severity of mitochondrial dysfunction.

Since patients are suspected of having sepsis with hypoperfusion (1. Blood lactate > 4 mmol/L, 2. Refractory hypotension: after bolus fluid 20 mL/kg and Systolic Blood Pressure still < 90 mmHg or require vasopressor), the sepsis bundle care will be started in the emergency department. The goals of this treatment are 1. A mean arterial pressure of > 65 is achieved by fluid resuscitation and vasopressor, 2. Lactate > 4 mmol/L or ScvO2 > 70 is achieved. After 6 hours following the beginning of resuscitation, blood examination for mitochondrial function, ScvO2 and ∆PCO2 will be determined. The correlation between these physiologic/biomarkers and mitochondrial function will be evaluated.

Aim #3 To investigate the roles of steroid administration on mitochondrial function in sepsis patients (Therapeutic trial) Aim 3.1 To investigate the therapeutic efficacy of steroids on the improvement mitochondrial function in sepsis patients Hypothesis: Steroids administration improve mitochondrial function in norepinephrine-resistant sepsis.

After resuscitation, hypoperfusion in the sepsis patients will be treated by fluid resuscitation and vasopressor. Some groups of patients may be not responsive to this treatment (MAP <65 mmHg), administration of steroids to this group will be blindly randomized (treatment and control group). During resuscitation of septic shock patients with fluid resuscitation and vasopressors, some may not respond to treatment (MAP < 65 mmHg). Patients who have shock refractory to fluid resuscitation and norepinephrine therapy for more than 0.5 mcg/kg/min will be blindly randomized to receive steroid (treatment group) or placebo (control group). Blood samples will be obtained to determine mitochondrial functioning before, at day 1 and day 7 after administration of study medications in both groups.

Aim 3.2. To investigate the efficacy of steroids on the reduction mortality rate in sepsis patients with norepinephrine-resistant hypotension Hypothesis: Steroids improve survival in septic shock patients with norepinephrine-resistant hypotension.

During resuscitation of septic shock patients with fluid resuscitation and vasopressors, some may not respond to treatment (MAP < 65 mmHg). Patients who have shock refractory to fluid resuscitation and norepinephrine administration more than 0.5 mcg/kg/min will be blindly randomized to receive steroid (treatment group) or placebo (control group). Blood samples will be obtained to determine mitochondrial functioning before, at day 1 and day 7 after administration of study medications in both groups. Thirty-day survival will be analyzed by a survival analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years of age)
2. Diagnosis of sepsis within 1 hour after presentation to the emergency department: known or presumed infection and SOFA score > 2 (table1)
3. Norepinephrine-resistant hypotension (refractory hypotension and not response to norepinephrine dose ≥ 0.5 mcg/k/min)

Exclusion Criteria:

1. Known pregnancy
2. Primary diagnosis of:

   1. acute cerebral vascular event
   2. acute coronary syndrome
   3. acute cardiogenic pulmonary edema
   4. status asthmaticus
   5. major cardiac arrhythmia (as part of primary diagnosis)
   6. seizure
   7. drug overdose
   8. injury from burn or trauma
3. Hemodynamic instability due to active hemorrhage
4. Requirement for immediate surgery
5. Do-Not-Attempt-Resuscitation (DNAR) order
6. Advanced directives restricting implementation of the resuscitation protocol
7. Transferred from another in-hospital setting
8. Sepsis or septic shock is not final diagnosis
9. Known history of HIV infection with suspected or known Cluster of differentiation 4 (CD4) <100 /mm2
10. Contraindication to central venous catheterization
11. Contraindication to blood transfusion
12. Attending clinician deems aggressive resuscitation unsuitable
13. Known history of HIV infection with suspected or known CD4 <100 /mm2
14. Neurodegenerative disease (effected mitochondria function)
15. known case adrenal insufficiency or chronic steroid user (Patient in this group should receive Hydrocortisone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
To investigate the level of mitochondrial respiration after steroid administration | 7 days
  Mean level comparative of mitochondrial respiration* in "Hydrocortisone" and "No intervention" groups will be investigated at before, day 1 after and day 7 after administration of intervention.
  *Mitochondrial function are mitochondrial respiration (Oxygen consumption rate in basal respiration, adenosine triphosphate (ATP) production, maximal respiration, spare capacity, proton leak, and non-mitochondrial respiration; Report in picomole/min)
To investigate the level of mitochondrial stress after steroid administration | 7 days
  Mean level comparative of mitochondrial stress* in "Hydrocortisone" and "No intervention" groups will be investigated at before, day 1 after and day 7 after administration of intervention.
  *Mitochondrial stress (mass of superoxide per mitochondrial mass) and oxidative phosphorylation in each complex (densitometric analysis by western blot)
To evaluate survival in septic patients who have refractory shock after steroid administration | 28 days
  Evaluate survival comparison in "Hydrocortisone" and "No intervention" groups. In 28 days survival and survival analysis until 28 day.

SECONDARY OUTCOMES:
To investigate risk factor (Age, underlying disease, number of organ dysfunction) correlation with the mitochondrial function in sepsis patients | since emergency department admission until blood examination was collected, up to 24 hours.
  Since there are many suspected cases of sepsis in the emergency department, mitochondrial function* measurements will be collected. Additionally, the correlation among sex, age, obesity, underlying symptoms, cause of infection, pathogen, onset of fever before emergency department (ED) visit. Correlation between mitochondrial function and each factor will be compare in percent, mean or median in each group.
  *Mitochondrial function are mitochondrial respiration (Oxygen consumption rate in basal respiration, ATP production, maximal respiration, spare capacity, proton leak, and non-mitochondrial respiration), mitochondrial stress (mass of superoxide per mitochondrial mass) and oxidative phosphorylation in each complex (densitometric analysis by western blot)
To investigate severity level of sepsis (SOFA Score) correlation with the mitochondrial function in sepsis patients | since emergency department admission until blood examination was collected, up to 24 hours.
  Since there are many suspected cases of sepsis in the emergency department, mitochondrial function* measurements will be collected. SOFA score**when patient visiting ED. Correlation between mitochondrial function and SOFA score present in linear correlation.
  *Mitochondrial function are mitochondrial respiration (Oxygen consumption rate in basal respiration, ATP production, maximal respiration, spare capacity, proton leak, and non-mitochondrial respiration), mitochondrial stress (mass of superoxide per mitochondrial mass) and oxidative phosphorylation in each complex (densitometric analysis by western blot)
  **Sepsis-related organ failure assessment score, is used to track a person's status to determine the extent of a person's organ function. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Score range from 0 to 20, if SOFA score increase at least 2 points, sepsis will be diagnosis.
To investigate the association of level of mitochondrial function in sepsis with central venous oxygen saturation (ScvO2) | since emergency department admission until patient disposition form emergency department, up to 24 hours.
  The correlation between these physiologic/biomarkers and mitochondrial function* will be evaluated. ScvO2 separated in low, normal and high group (<70%, 70-80%, >80%). Each ScvO2 group calculate mitochondrial function in mean and analysis mean difference.
  *Mitochondrial function are mitochondrial respiration (Oxygen consumption rate in basal respiration, ATP production, maximal respiration, spare capacity, proton leak, and non-mitochondrial respiration), mitochondrial stress (mass of superoxide per mitochondrial mass) and oxidative phosphorylation in each complex (densitometric analysis by western blot)
To investigate the association of level of mitochondrial function in sepsis with serum lactate. | since emergency department admission until patient disposition form emergency department, up to 24 hours.
  The correlation between these physiologic/biomarkers and mitochondrial function* will be evaluated. Serum lactate separated in normal and high group (<2 mmol/L and >=2 mmol/L), . Each serum lactate group calculate mitochondrial function in mean and analysis mean difference.
  *Mitochondrial function are mitochondrial respiration (Oxygen consumption rate in basal respiration, ATP production, maximal respiration, spare capacity, proton leak, and non-mitochondrial respiration), mitochondrial stress (mass of superoxide per mitochondrial mass) and oxidative phosphorylation in each complex (densitometric analysis by western blot)
To investigate the association of level of mitochondrial function in sepsis with venous-to-arterial carbon dioxide tension difference (delta PCO2). | since emergency department admission until patient disposition form emergency department, up to 24 hours.
  The correlation between these physiologic/biomarkers and mitochondrial function* will be evaluated. Delta PCO2 in normal and high group (<6 mmHg, >=6mmHg). Each group of Delta PCO2 calculate mitochondrial function in mean and analysis mean difference.
  *Mitochondrial function are mitochondrial respiration (Oxygen consumption rate in basal respiration, ATP production, maximal respiration, spare capacity, proton leak, and non-mitochondrial respiration), mitochondrial stress (mass of superoxide per mitochondrial mass) and oxidative phosphorylation in each complex (densitometric analysis by western blot)

CONTACTS AND LOCATIONS:
Overall Officials: BORWON WITTAYACHAMNANKUL, MD, Principal Investigator — Emergency Department, Medicine Faculty, Chiang Mai University, Thailand
Locations (1):
- Emergency Department, Faculty of Medicine, Chaing Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No